CLINICAL TRIAL: NCT02813798
Title: A PHASE 1, NON-RANDOMIZED, OPEN-LABEL, SINGLE DOSE STUDY TO EVALUATE THE EFFECT OF RENAL IMPAIRMENT ON THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF RIVIPANSEL (PF-06460031) IN SUBJECTS WITH RENAL IMPAIRMENT AND IN HEALTHY SUBJECTS
Brief Title: A Study to Evaluate the Effect of IV Doses of Rivipansel on Subjects With Renal Impairment and in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B5201005
Record Dates: First submitted 2016-06-15; First posted 2016-06-27 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Renal Impairment; Healthy
Keywords: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — rivipansel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Mild Renal Impairment (Experimental): A single dose of IV Rivipansel over 20 minutes
  Interventions: Drug: Rivipansel
- Moderate Renal Impairment (Experimental): A single dose of IV Rivipansel over 20 minutes
  Interventions: Drug: Rivipansel
- Severe Renal Impairment (Experimental): A single dose of IV Rivipansel over 20 minutes
  Interventions: Drug: Rivipansel
- Normal Renal Functions (Experimental): A single dose of IV Rivipansel over 20 minutes
  Interventions: Drug: Rivipansel

INTERVENTIONS:
Drug: Rivipansel — A single 840mg dose of Rivipansel over 20 minutes
  Other Names: GMI-1070

SUMMARY:
The purpose of this study is to determine the effect of renal impairment on rivipansel.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of non-childbearing potential or male subjects
* Body Mass Index (BMI) of 17.5 to 40.0 kg/m2
* Stable renal function

Exclusion Criteria:

* A positive urine drug screen for illicit drugs
* Treatment with an investigational drug within 30 days of the dose of study medication
* Pregnant females, breastfeeding female subjects and male subjects with partners currently pregnant
* Use of herbal supplements in the 28 days prior to the dose of study medication
* Blood donation (excluding plasma donation) of approximately 1 pint or more within 56 days prior to study medication
* Requiring dialysis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 to infinity or area under the concentration-time curve from time 0 to the time of the last quantifiable concentration, as data permit | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72 and 96 H following single dose administration
Clearance (CL) | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72 and 96 H following single dose administration
Renal clearance | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72 and 96 H following single dose administration
Physical examination | Baseline up to 96 hours
Assessment of adverse events | Baseline up to 28 days
Assessment of 12-lead electrocardiograms | Baseline up to 96 hours
Assessment of vital signs | Baseline up to 96 hours
Assessment of laboratory tests | Baseline up to 96 hours

SECONDARY OUTCOMES:
Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72 and 96 H following single dose administration
Peak or maximum observed concentration | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72 and 96 H following single dose administration
Time to reach maximum concentration | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72 and 96 H following single dose administration
Terminal half life | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72 and 96 H following single dose administration
Apparent volume of distribution | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72 and 96 H following single dose administration
Amount of unchanged drug excreted into urine over 96 hours | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72 and 96 H following single dose administration
Percentage of dose excreted unchanged into urine over 96 hours | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72 and 96 H following single dose administration
Fraction of unbound | Samples are collected pre-dose and at 0.33, 1, 3, 6, 8, 12, 16, 24, 36, 48, 72 and 96 H following single dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tammara BK, Ryan K, Plotka A, Shafer FE, Wei H, Readett D, Fang A, Korth-Bradley JM. Effect of Renal or Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of Intravenous Rivipansel. Clin Pharmacol Drug Dev. 2020 Nov;9(8):918-928. doi: 10.1002/cpdd.842. Epub 2020 Jun 24. PMID 32579796